CLINICAL TRIAL: NCT00339183
Title: A Randomized, Multicenter Phase 3 Study to Compare the Efficacy of Panitumumab in Combination With Chemotherapy to the Efficacy of Chemotherapy Alone in Patients With Previously Treated Metastatic Colorectal Cancer
Brief Title: Comparison of Treatment Effect of Chemotherapy With Panitumumab to Chemotherapy Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20050181
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Results first posted 2014-05-06 (Estimated); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Oncology; Cancer; Metastatic Colorectal Cancer; EGFr; Panitumumab; Clinical Trial; Amgen
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Panitumumab; IFL protocol

ARMS (2):
- Panitumumab Plus FOLFIRI (Experimental): Participants received panitumumab as an intravenous (IV) infusion at a dose of 6 mg/kg plus a standard chemotherapy regimen (FOLFIRI) consisting of 5-fluorouracil (5-FU), leucovorin and irinotecan. Treatment was administered in cycles every two weeks.
  Interventions: Drug: Panitumumab; Drug: FOLFIRI
- FOLFIRI Alone (Active Comparator): Participants received standard chemotherapy regimen (FOLFIRI) consisting of 5-FU, leucovorin and irinotecan. Treatment is administered in cycles every two weeks.
  Interventions: Drug: FOLFIRI

INTERVENTIONS:
Drug: Panitumumab — Panitumumab was administered by IV infusion on Day 1 of each 14-day cycle, just before administration of FOLFIRI chemotherapy.
  Other Names: Vectibix®
  Arms: Panitumumab Plus FOLFIRI
Drug: FOLFIRI — FOLFIRI chemotherapy was initiated on Day 1 of each treatment cycle at the following starting doses: irinotecan 180 mg/m^2, leucovorin 400 mg/m^2 racemate (or 200 mg/m^2 I-leucovorin), 5-FU bolus 400 mg/m^2, 5-FU infusion 2400 mg/m^2.

SUMMARY:
The purpose of this study is to evaluate the treatment effect of panitumumab plus FOLFIRI compared to FOLFIRI alone as second line therapy for metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman at least 18 years old
* Diagnosis of metastatic colorectal cancer (mCRC)
* One and only one chemotherapy regimen for mCRC consisting of first-line 5-FU -based chemotherapy
* Radiologically documented disease progression per modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria during treatment or within 6 months of last dose of first-line chemotherapy
* At least 1 uni-dimensionally measurable lesion of at least 20 mm per modified RECIST
* Eastern Cooperative Oncology Group (ECOG) status of 0, 1, or 2
* Paraffin-embedded tumor tissue from the primary tumor or metastasis available for central analyses
* Adequate hematologic, renal, and hepatic functions
* Negative pregnancy test within 72 hours of enrollment
* Other protocol-specified criteria may apply

Exclusion Criteria:

* History of or known presence of central nervous system (CNS) metastases
* History of another primary cancer within 5 years of randomization
* Prior irinotecan therapy
* Prior anti-epidermal growth factor receptor (EGFr) antibody therapy or treatment with small molecule EGFr inhibitors
* Any investigational agent or therapy within 30 days before randomization
* Known allergy or hypersensitivity to irinotecan, 5-FU or leucovorin
* History of interstitial lung disease or evidence of interstitial lung disease on baseline chest computed tomography (CT) scan
* Active inflammatory bowel disease or other bowel disease causing chronic diarrhea
* Known positive tests for human immunodefiency virus (HIV), hepatitis C viris (HCV), acute or chronic active hepatitis B virus (HBV)
* Major surgery within 28 days of randomization or minor surgical procedure within 14 days of randomization
* Pregnant or breast-feeding
* Man or woman of child-bearing potential not consenting to use adequate contraceptive methods or abstinence during the course of the study and for 6 months after last study drug administration (women) or 1 month after last study drug administration (men)
* Other protocol-specified criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1186 (Actual)
Dates: Start 2006-06-30 (Actual); Primary Completion 2009-04-01 (Actual); Study Completion 2010-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Peeters M, Price TJ, Cervantes A, Sobrero AF, Ducreux M, Hotko Y, Andre T, Chan E, Lordick F, Punt CJ, Strickland AH, Wilson G, Ciuleanu TE, Roman L, Van Cutsem E, Tian Y, Sidhu R. Final results from a randomized phase 3 study of FOLFIRI +/- panitumumab for second-line treatment of metastatic colorectal cancer. Ann Oncol. 2014 Jan;25(1):107-16. doi: 10.1093/annonc/mdt523. PMID 24356622
- [Background] Peeters M, Price TJ, Cervantes A, Sobrero AF, Ducreux M, Hotko Y, Andre T, Chan E, Lordick F, Punt CJ, Strickland AH, Wilson G, Ciuleanu TE, Roman L, Van Cutsem E, Tzekova V, Collins S, Oliner KS, Rong A, Gansert J. Randomized phase III study of panitumumab with fluorouracil, leucovorin, and irinotecan (FOLFIRI) compared with FOLFIRI alone as second-line treatment in patients with metastatic colorectal cancer. J Clin Oncol. 2010 Nov 1;28(31):4706-13. doi: 10.1200/JCO.2009.27.6055. Epub 2010 Oct 4. PMID 20921462
- [Background] Author and team decided to wait for CALGB RAS data presented Sept 29 at ESMO.
- [Background] Peeters M, Price T, Taieb J, Geissler M, Rivera F, Canon JL, Pentheroudakis G, Koukakis R, Burdon P, Siena S. Relationships between tumour response and primary tumour location, and predictors of long-term survival, in patients with RAS wild-type metastatic colorectal cancer receiving first-line panitumumab therapy: retrospective analyses of the PRIME and PEAK clinical trials. Br J Cancer. 2018 Aug;119(3):303-312. doi: 10.1038/s41416-018-0165-z. Epub 2018 Jul 17. PMID 30013091
- [Derived] Shi Y, Wan X, Tan C, Li J, Peng L. Model-Based Cost-Effectiveness Analysis of Panitumumab Plus FOLFIRI for the Second-Line Treatment of Patients with Wild-Type Ras Metastatic Colorectal Cancer. Adv Ther. 2020 Feb;37(2):847-859. doi: 10.1007/s12325-019-01214-y. Epub 2020 Jan 4. PMID 31902066
- [Derived] Boeckx N, Koukakis R, Op de Beeck K, Rolfo C, Van Camp G, Siena S, Tabernero J, Douillard JY, Andre T, Peeters M. Effect of Primary Tumor Location on Second- or Later-line Treatment Outcomes in Patients With RAS Wild-type Metastatic Colorectal Cancer and All Treatment Lines in Patients With RAS Mutations in Four Randomized Panitumumab Studies. Clin Colorectal Cancer. 2018 Sep;17(3):170-178.e3. doi: 10.1016/j.clcc.2018.03.005. Epub 2018 Mar 8. PMID 29627309
- [Derived] Peeters M, Oliner KS, Price TJ, Cervantes A, Sobrero AF, Ducreux M, Hotko Y, Andre T, Chan E, Lordick F, Punt CJ, Strickland AH, Wilson G, Ciuleanu TE, Roman L, Van Cutsem E, He P, Yu H, Koukakis R, Terwey JH, Jung AS, Sidhu R, Patterson SD. Analysis of KRAS/NRAS Mutations in a Phase III Study of Panitumumab with FOLFIRI Compared with FOLFIRI Alone as Second-line Treatment for Metastatic Colorectal Cancer. Clin Cancer Res. 2015 Dec 15;21(24):5469-79. doi: 10.1158/1078-0432.CCR-15-0526. Epub 2015 Sep 4. PMID 26341920
- [Derived] Peeters M, Kafatos G, Taylor A, Gastanaga VM, Oliner KS, Hechmati G, Terwey JH, van Krieken JH. Prevalence of RAS mutations and individual variation patterns among patients with metastatic colorectal cancer: A pooled analysis of randomised controlled trials. Eur J Cancer. 2015 Sep;51(13):1704-13. doi: 10.1016/j.ejca.2015.05.017. Epub 2015 Jun 3. PMID 26049686
- [Derived] Weeraratne D, Chen A, Pennucci JJ, Wu CY, Zhang K, Wright J, Perez-Ruixo JJ, Yang BB, Kaliyaperumal A, Gupta S, Swanson SJ, Chirmule N, Starcevic M. Immunogenicity of panitumumab in combination chemotherapy clinical trials. BMC Clin Pharmacol. 2011 Nov 9;11:17. doi: 10.1186/1472-6904-11-17. PMID 22070868
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 30 June 2006; Last patient enrolled 13 March 2008.
Groups:
- Panitumumab Plus FOLFIRI: Participants were randomized to 6 mg/kg panitumumab intravenous infusion plus a standard chemotherapy regimen (FOLFIRI) consisting of 5-FU, leucovorin and irinotecan. Treatment was administered in cycles every two weeks.
- FOLFIRI Alone: Participants were randomized to receive a standard chemotherapy regimen (FOLFIRI) consisting of 5-FU, leucovorin and irinotecan. Treatment was administered in cycles every two weeks.
Period: Overall Study
Arm/Group | Panitumumab Plus FOLFIRI | FOLFIRI Alone
Started | 591 | 595
Received Study Drug | 588 (Includes one participant who received FOLFIRI Alone) | 593
Completed | 470 (Indicates participants who had completed the safety visit 30 days after last dose or had died) | 490 (Indicates participants who had completed the safety visit 30 days after last dose or had died)
Not Completed | 121 | 105
Not completed — Adverse Event | 5 | 3
Not completed — Withdrawal by Subject | 16 | 19
Not completed — Physician Decision | 2 | 4
Not completed — Lost to Follow-up | 17 | 17
Not completed — Protocol-specified criteria | 12 | 8
Not completed — Missing reason | 3 | 1
Not completed — Other | 46 | 40
Not completed — Ongoing | 20 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panitumumab Plus FOLFIRI | FOLFIRI Alone | Total
Number analyzed (Participants) | 591 | 595 | 1186
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (10.5) | 60.9 (10.6) | 60.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245 | 219 | 464
  Male | 346 | 376 | 722
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 568 | 569 | 1137
  Black or African American | 4 | 5 | 9
  Hispanic or Latino | 2 | 3 | 5
  Asian | 2 | 3 | 5
  Japanese | 9 | 11 | 20
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Aborigine | 2 | 1 | 3
  Other | 3 | 2 | 5
KRAS Status [Number; unit: participants] — KRAS, the human homolog of the Kirsten rat sarcoma-2 virus oncogene
  participants
    Wild-type KRAS | 303 | 294 | 597
    Mutant KRAS | 238 | 248 | 486
    Unevaluable KRAS | 50 | 53 | 103
Prior Oxaliplatin Exposure for mCRC [Number; unit: participants] — mCRC: metastatic colorectal cancer
  participants
    No | 179 | 182 | 361
    Yes | 412 | 413 | 825
Prior Bevacizumab Exposure for mCRC [Number; unit: participants]
  No | 480 | 483 | 963
  Yes | 111 | 112 | 223
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; Grade 2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours; Grade 3: Capable of only limited self care, confined to a bed or chair > 50% of waking hours; Grade 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; Grade 5: Dead
  participants
    Grade 0 or 1 | 564 | 565 | 1129
    Grade 2 | 27 | 30 | 57

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was defined as the time from randomization to first disease progression per modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria or death, based on independent central radiological assessment. Participants who were alive but did not meet criteria for progression by the data cutoff date were censored at their last evaluable disease assessment date.
  Progressive disease is defined as a ≥ 20% increase in the size of target lesions or unequivocal progression of existing non-target lesions or any new lesions.
Time Frame: From randomization until the data cut-off date of 8 April 2008. Maximum follow-up time was 17 months.
Population: KRAS Efficacy Analysis Set (participants for whom KRAS status was assessed)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Wild-type KRAS - Panitumumab Plus FOLFIRI: Participants with wild-type KRAS were randomized to 6 mg/kg panitumumab plus FOLFIRI chemotherapy regimen administered in cycles every two weeks.
- Wild-type KRAS - FOLFIRI Alone: Participants with wild-type KRAS were randomized to FOLFIRI chemotherapy regimen administered in cycles every two weeks.
- Mutant KRAS - Panitumumab Plus FOLFIRI: Participants with mutant KRAS were randomized to 6 mg/kg panitumumab plus FOLFIRI chemotherapy regimen administered in cycles every two weeks.
- Mutant KRAS - FOLFIRI Alone: Participants with mutant KRAS were randomized to FOLFIRI chemotherapy regimen administered in cycles every two weeks.
Arm/Group | Wild-type KRAS - Panitumumab Plus FOLFIRI | Wild-type KRAS - FOLFIRI Alone | Mutant KRAS - Panitumumab Plus FOLFIRI | Mutant KRAS - FOLFIRI Alone
Number analyzed (Participants) | 303 | 294 | 238 | 248
months | 5.9 [5.5 to 6.7] | 3.9 [3.7 to 5.3] | 5.0 [3.8 to 5.6] | 4.9 [3.6 to 5.6]
Statistical Analysis 1: Comparison: Wild-type KRAS - Panitumumab Plus FOLFIRI vs Wild-type KRAS - FOLFIRI Alone; An overall 5% significance level was used to compare treatments with respect to both overall survival (OS) and PFS. A 4% and 1% level (2-sided) was used to independently test OS and PFS, respectively; Test type: Superiority or Other; p = 0.0036, Stratified log-rank test; P-value based on a 2-sided log-rank test stratified by ECOG (0 or 1 vs. 2), prior bevacizumab exposure, and prior oxaliplatin exposure (yes or no); Normal score = -2.91 — A normal score <0 indicates fewer than expected events for the Panitumumab plus FOLFIRI arm and therefore a longer progression-free survival time
Statistical Analysis 2: Comparison: Mutant KRAS - Panitumumab Plus FOLFIRI vs Mutant KRAS - FOLFIRI Alone; PFS in the Mutant Efficacy Analysis Set was compared at a 1% level conditional upon first demonstrating a significant difference in PFS in the Wild-type KRAS Efficacy Analysis Set; Test type: Superiority or Other; p = 0.1448, Stratified log-rank test; P-value based on a 2-sided log-rank test stratified by ECOG (0 or 1 vs. 2), prior bevacizumab exposure and prior oxaliplatin exposure (yes or no); Normal score = -1.46 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization to the date of death. Participants who had not died by the analysis data cutoff date had their time of death censored at their last contact date.
Time Frame: From randomization until the data cut-off date of 30 April 2009. Maximum follow-up time was 33 months
Population: KRAS Efficacy Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Wild-type KRAS - Panitumumab Plus FOLFIRI | Wild-type KRAS - FOLFIRI Alone | Mutant KRAS - Panitumumab Plus FOLFIRI | Mutant KRAS - FOLFIRI Alone
Number analyzed (Participants) | 303 | 294 | 238 | 248
months | 14.5 [13.0 to 16.0] | 12.5 [11.2 to 14.2] | 11.8 [10.4 to 13.3] | 11.1 [10.3 to 12.4]
Statistical Analysis 1: Comparison: Wild-type KRAS - Panitumumab Plus FOLFIRI vs Wild-type KRAS - FOLFIRI Alone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1154, Stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Normal score = -1.57 — A normal score <0 indicates fewer than expected events for the Panitumumab plus FOLFIRI arm and therefore a longer overall survival time
Statistical Analysis 2: Comparison: Mutant KRAS - Panitumumab Plus FOLFIRI vs Mutant KRAS - FOLFIRI Alone; The treatment effect on OS in the Mutant KRAS Efficacy Analysis Set was compared at the 4% level conditional on first demonstrating a significant OS treatment effect in the Wild-type KRAS Efficacy Analysis Set; Test type: Superiority or Other; p = 0.5503, Stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Normal score = -0.60 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Participants With an Objective Response
Description: Participants were evaluated for tumor response per the modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria every 8 weeks until disease progression. Objective response was defined as the incidence of either a confirmed complete or partial response (CR or PR) while on study, as determined by blinded independent central review and confirmed no less than 4-weeks after the criteria for response are first met. CR: Disappearance of all target and non-target lesions and no new lesions. PR: At least a 30% decrease in the sum of the longest diameter of target lesions and no progression of non-target or no new lesions, or, disappearance of all target lesions and the persistence of ≥ 1 non-target lesion not qualifying for either CR or progressive disease. Participants without a post-baseline assessment were considered non-responders.
Time Frame: Every 8 weeks until disease progression up to the data cut-off date of 30 April 2009. Maximum time on follow-up was 33 months.
Population: KRAS Central Tumor Response Analysis Set: subset of participants with at least one uni-dimensionally measurable lesion per the modified RECIST criteria per blinded central radiology review for whom KRAS was assessed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Wild-type KRAS - Panitumumab Plus FOLFIRI | Wild-type KRAS - FOLFIRI Alone | Mutant KRAS - Panitumumab Plus FOLFIRI | Mutant KRAS - FOLFIRI Alone
Number analyzed (Participants) | 297 | 285 | 232 | 237
percentage of participants | 35.35 [29.92 to 41.08] | 9.82 [6.63 to 13.89] | 13.36 [9.26 to 18.43] | 13.92 [9.78 to 19.00]
Statistical Analysis 1: Comparison: Wild-type KRAS - Panitumumab Plus FOLFIRI vs Wild-type KRAS - FOLFIRI Alone; Test type: Superiority or Other; p < 0.0001, Stratified exact test; Adjusted for ECOG score, prior bevacizumab exposure, prior oxaliplatin exposure; Odds Ratio (OR) = 5.33, 95% CI 2-sided [3.21 to 8.60] — The odds ratio is defined as the odds of having an objective response in the panitumumab plus arm relative to the odds on the FOLFIRI alone arm
Statistical Analysis 2: Comparison: Mutant KRAS - Panitumumab Plus FOLFIRI vs Mutant KRAS - FOLFIRI Alone; Test type: Superiority or Other; p = 1.0000, Stratified exact test; Adjusted for ECOG score, prior bevacizumab exposure, prior oxaliplatin exposure; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.56 to 1.76] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Time to Disease Progression
Description: Time to progression was defined as the time from the randomization date to the date of first observed disease progression per the modified RECIST criteria. Participants not meeting these criteria by the analysis data cutoff date were censored at their last evaluable disease assessment date.
  Progressive disease is defined as a ≥ 20% increase in the size of target lesions or unequivocal progression of existing non-target lesions or any new lesions.
Time Frame: From randomization until the data cut-off date of 30 April 2009. Maximum follow-up time was 33 months
Population: KRAS Efficacy Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Wild-type KRAS - Panitumumab Plus FOLFIRI | Wild-type KRAS - FOLFIRI Alone | Mutant KRAS - Panitumumab Plus FOLFIRI | Mutant KRAS - FOLFIRI Alone
Number analyzed (Participants) | 303 | 294 | 238 | 248
months | 7.3 [5.9 to 7.5] | 5.3 [3.9 to 5.7] | 5.5 [4.5 to 5.7] | 5.5 [4.2 to 5.7]

5. Secondary Outcome: Duration of Response
Description: Calculated only for those participants with an objective response as the time from the first objective response (subsequently confirmed within no less than 4 weeks) to first observed disease progression per modified-RECIST criteria. Participants not meeting these criteria by the analysis data cutoff date were censored at their last evaluable disease assessment date.
  Progressive disease is defined as a ≥ 20% increase in the size of target lesions or unequivocal progression of existing non-target lesions or any new lesions.
Time Frame: From randomization until the data cut-off date of 30 April 2009. Maximum follow-up time was 33 months
Population: KRAS Central Tumor Response Analysis Set: Responders
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Wild-type KRAS - Panitumumab Plus FOLFIRI | Wild-type KRAS - FOLFIRI Alone | Mutant KRAS - Panitumumab Plus FOLFIRI | Mutant KRAS - FOLFIRI Alone
Number analyzed (Participants) | 105 | 28 | 31 | 33
months | 7.6 [6.7 to 9.4] | 6.6 [5.7 to 10.4] | 6.0 [5.4 to 7.4] | 7.4 [4.0 to 8.1]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: A serious adverse event (SAE) is defined by regulatory authorities as one that • is fatal • is life threatening (places the subject at immediate risk of death) • requires in-patient hospitalization or prolongation of existing hospitalization • results in persistent or significant disability/incapacity • is a congenital anomaly/birth defect • other significant medical hazard. The relationship of the adverse event to the study treatment was assessed by the Investigator by means of the question: "Is there a reasonable possibility that the event may have been caused by the study treatment?"
Time Frame: From randomization until the data cut-off date of 30 April 2009. Maximum follow-up time was 33 months.
Population: Safety analysis set: all participants who received at least 1 dose of panitumumab or chemotherapy. One participant was randomized to Panitumumab Plus FOLFIRI, but received FOLFIRI Alone and is included in the FOLFIRI Alone group for safety analyses.
Measure: Number; unit: participants
Groups:
- Panitumumab Plus FOLFIRI: Participants received 6 mg/kg panitumumab IV plus a standard chemotherapy regimen (FOLFIRI) consisting of 5-FU, leucovorin and irinotecan. Treatment was administered in cycles every two weeks.
- FOLFIRI Alone: Participants received FOLFIRI chemotherapy regimen administered in cycles every two weeks.
Arm/Group | Panitumumab Plus FOLFIRI | FOLFIRI Alone
Number analyzed (Participants) | 587 | 594
participants
  Any adverse event | 584 | 573
  Serious adverse event | 232 | 175
  Leading to discontinuation of any study drug | 123 | 64
  Treatment-related adverse event (TRAE) | 577 | 542
  Serious treatment-related adverse event | 124 | 90
  TRAE leading to discontinuation of any study drug | 97 | 34

ADVERSE EVENTS:
Time Frame: The median treatment period was approximately 6.2 months in the Panitumumab plus FOLFIRI arm, and 4.7 months in the FOLFIRI Alone arm.
Description: One participant was randomized to Panitumumab Plus FOLFIRI, but received FOLFIRI Alone and is included in the FOLFIRI Alone group for safety analyses.
  The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Panitumumab Plus FOLFIRI | FOLFIRI Alone
Serious Adverse Events (participants affected / at risk) | 232/587 | 175/594
Other Adverse Events (participants affected / at risk) | 575/587 | 546/594
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus FOLFIRI (N=587) | FOLFIRI Alone (N=594)
Anaemia (Blood and lymphatic system disorders) | 5 | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 11 | 16
Leukopenia (Blood and lymphatic system disorders) | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 12
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 2
Aplasia (Congenital, familial and genetic disorders) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 12 | 13
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 1 | 0
Anorectal disorder (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 3
Colitis (Gastrointestinal disorders) | 1 | 1
Colonic obstruction (Gastrointestinal disorders) | 2 | 4
Colonic stenosis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 33 | 23
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Faecal vomiting (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 2
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Ileal perforation (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 4 | 4
Intestinal obstruction (Gastrointestinal disorders) | 9 | 9
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 12 | 5
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Sigmoiditis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 6 | 4
Stomatitis (Gastrointestinal disorders) | 1 | 3
Subileus (Gastrointestinal disorders) | 2 | 4
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 17 | 13
Accidental death (General disorders) | 1 | 0
Asthenia (General disorders) | 8 | 1
Catheter related complication (General disorders) | 2 | 0
Catheter site related reaction (General disorders) | 1 | 0
Catheter thrombosis (General disorders) | 1 | 1
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 3 | 3
Chills (General disorders) | 1 | 2
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 5 | 5
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 6 | 8
Generalised oedema (General disorders) | 1 | 0
Hyperthermia (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 2
Mucosal inflammation (General disorders) | 2 | 4
Multi-organ failure (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 7 | 1
Performance status decreased (General disorders) | 4 | 0
Pyrexia (General disorders) | 24 | 16
Sudden death (General disorders) | 2 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 1 | 0
Cholangiolitis (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 3
Cholestasis (Hepatobiliary disorders) | 2 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 2
Abdominal infection (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Actinomycotic pulmonary infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 1
Biliary sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Campylobacter infection (Infections and infestations) | 1 | 0
Candida sepsis (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 7 | 3
Catheter sepsis (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 6 | 1
Device related infection (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 3 | 1
Influenza (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 1
Oropharyngitis fungal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 4
Post procedural infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 4 | 3
Septic shock (Infections and infestations) | 1 | 2
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 2 | 0
Subcutaneous abscess (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 5 | 3
Urosepsis (Infections and infestations) | 2 | 1
Vaginitis bacterial (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 1
Drug administration error (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Perinephric collection (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 0 | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
General physical condition abnormal (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 2 | 0
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 20 | 11
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hip swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 10
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour local invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 2 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 3
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1
Cholinergic syndrome (Nervous system disorders) | 1 | 1
Chorea (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Epiduritis (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 2
Nervous system disorder (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 1
Status epilepticus (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Renal colic (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 2
Renal failure acute (Renal and urinary disorders) | 3 | 3
Ureteric obstruction (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Genital ulceration (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Perineal fistula (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 17 | 10
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 3 | 0
Liver operation (Surgical and medical procedures) | 0 | 1
Stent placement (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 7 | 2
Embolism (Vascular disorders) | 0 | 1
Embolism venous (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 4 | 2
Vena cava thrombosis (Vascular disorders) | 1 | 1
Venous thrombosis (Vascular disorders) | 1 | 2
Venous thrombosis limb (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus FOLFIRI (N=587) | FOLFIRI Alone (N=594)
Anaemia (Blood and lymphatic system disorders) | 79 | 110
Leukopenia (Blood and lymphatic system disorders) | 64 | 60
Neutropenia (Blood and lymphatic system disorders) | 207 | 209
Thrombocytopenia (Blood and lymphatic system disorders) | 20 | 39
Conjunctivitis (Eye disorders) | 81 | 11
Abdominal pain (Gastrointestinal disorders) | 122 | 105
Abdominal pain upper (Gastrointestinal disorders) | 37 | 33
Constipation (Gastrointestinal disorders) | 139 | 125
Diarrhoea (Gastrointestinal disorders) | 372 | 321
Dry mouth (Gastrointestinal disorders) | 30 | 10
Dyspepsia (Gastrointestinal disorders) | 40 | 32
Nausea (Gastrointestinal disorders) | 276 | 269
Stomatitis (Gastrointestinal disorders) | 131 | 75
Vomiting (Gastrointestinal disorders) | 154 | 162
Asthenia (General disorders) | 74 | 81
Fatigue (General disorders) | 203 | 186
Mucosal inflammation (General disorders) | 121 | 68
Oedema peripheral (General disorders) | 59 | 41
Pain (General disorders) | 43 | 29
Pyrexia (General disorders) | 105 | 89
Paronychia (Infections and infestations) | 102 | 3
Weight decreased (Investigations) | 60 | 29
Anorexia (Metabolism and nutrition disorders) | 146 | 93
Hypocalcaemia (Metabolism and nutrition disorders) | 32 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 65 | 27
Hypomagnesaemia (Metabolism and nutrition disorders) | 120 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 62 | 44
Dizziness (Nervous system disorders) | 36 | 35
Headache (Nervous system disorders) | 34 | 40
Insomnia (Psychiatric disorders) | 53 | 48
Cough (Respiratory, thoracic and mediastinal disorders) | 42 | 55
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 54 | 36
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 52 | 38
Acne (Skin and subcutaneous tissue disorders) | 80 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 124 | 136
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 141 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 129 | 23
Erythema (Skin and subcutaneous tissue disorders) | 92 | 16
Nail disorder (Skin and subcutaneous tissue disorders) | 43 | 8
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 54 | 22
Pruritus (Skin and subcutaneous tissue disorders) | 107 | 18
Rash (Skin and subcutaneous tissue disorders) | 330 | 38
Skin fissures (Skin and subcutaneous tissue disorders) | 94 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.